CLINICAL TRIAL: NCT03094169
Title: Phase 1a/2a Dose Escalation Trial to Determine Safety, Tolerance, MTD, and Preliminary Antineoplastic Activity of AVID100, in Patients With Advanced or Metastatic Solid Tumors of Epithelial Origin
Brief Title: AVID100 in Advanced Epithelial Carcinomas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Formation Biologics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVID100-01
Record Dates: First submitted 2017-02-06; First posted 2017-03-29 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2022-03

CONDITIONS: Solid Tumor, Adult; Triple Negative Breast Cancer; Head and Neck Squamous Cell Carcinoma; Non Small Cell Lung Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Uncontrolled, open label, non-randomized, Enrollment in the order of confirmation of eligibility, Escalating doses of study drug in sequential patient cohorts (Phase 1a). Uncontrolled, open label, non-randomised. Enrollment into three individual Phase 2a study cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose escalation (Experimental): Minimum of 1 to 3 patients per dose cohort; approximately 4 dose cohorts to be evaluated to establish the Maximum tolerated dose.
  Interventions: Drug: AVID100 IV
- Phase 2a Triple Negative Breast Cancer (Experimental): Addition of up to 15 patients in each of 2 subpopulations of patients with triple negative breast cancer (30 total). One group of 15 patients will have 3+ EGFR over-expression. The second group will have 2+ EGFR over-expression.
  Interventions: Drug: AVID100 IV
- Phase 2a Head and Neck Carcinoma (Experimental): Addition of 15 patients with squamous head and neck carcinoma. Patients will have 3+ EGFR over-expression.
  Interventions: Drug: AVID100 IV
- Phase 2a Non-Small Cell Lung Carcinoma (Experimental): Addition of 15 patients with squamous histology non-small cell lung carcinoma. Patients will have 3+ EGFR over-expression
  Interventions: Drug: AVID100 IV

INTERVENTIONS:
Drug: AVID100 IV — AVID100 is administered once every 3 weeks

SUMMARY:
Approximately 90 male and female patients with documented solid tumor malignancies of epithelial origin that are locally advanced or metastatic, and either refractory to standard therapy or for whom no standard therapy is available, will be entered into this Phase 1a/2a, multicenter, open-label, dose-escalation, cohort study of AVID100. Phase 2a will include evaluation of patient with EGFR-overexpressing squamous histology non-small cell lung cancer, squamous cell carcinoma of the head and neck, and triple negative breast cancer

DETAILED DESCRIPTION:
On Day 1 of study, patients will receive study drug administered by 2-hour IV infusion. AVID100 will be administered once every 3 weeks (Q3W) with administration on Day 1 of the first week, followed by a 3-week recovery period. In Phase 2a AVID100 will be administered at a dose of 220 mg/m2.

Evidence of progressive disease at any point in the study will necessitate withdrawal of the patient from further participation so that alternative management of their malignancy may be considered. All patients will be followed to further evaluate safety as well as evidence of the anti-tumor effects of AVID100 in these selected patient populations. If anti-tumor activity is observed additional patients may be added to the planned Phase 2a patient populations to further characterize these effects.

ELIGIBILITY:
Inclusion Criteria (Phase 1):

1. Patients with a documented (histologically- or cytologically-proven) solid tumor epithelial carcinoma that is locally advanced or metastatic
2. Patients with a malignancy that is either refractory to standard therapy, or for which no standard therapy is available
3. Patients with a malignancy that is currently not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor
4. Phase 1a Dose-Escalation Cohorts: Patients with measurable or non-measurable disease according to RECIST, v1.1 criteria. To include patients reasonably likely to express EGFR.

Inclusion Criteria (Phase 2a)

1. Patients with measurable disease according to RECIST, v1.1 criteria.
2. Patients with triple negative breast cancer who are either EGFR 2+ or EGFR 3+ by validated IHC assay.
3. Patients with squamous non-small cell lung cancer who are EGFR 3+ by validated IHC assay.
4. Patients with squamous cell carcinoma of the head and neck who are EGFR 3+ by validated IHC assay.
5. Patients whose malignancy is either refractory to standard therapy, or for which no standard therapy is available
6. Patients whose malignancy is currently not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor

Patients to be Excluded (patients must not meet any of the following criteria Phase 1 only)

1. Women who are pregnant or lactating. Women of child-bearing potential (WOCBP) and fertile men with WOCBP partner(s), not using and not willing to use a medically effective method of contraception.
2. Patients with known central nervous system (CNS) or leptomeningeal metastases, or spinal cord compression not controlled by prior surgery or radiotherapy, or patients with symptoms suggesting CNS involvement for which treatment is required
3. Patients with a malignancy other than that of epithelial origin
4. Patients with hematologic abnormalities at baseline
5. Patients with a significant cardiovascular disease or condition
6. Patients with a significant ocular disease or condition
7. Patients with a significant pulmonary disease or condition
8. History of pneumonia within 6 months prior to the first study drug administration
9. Patients with significant gastrointestinal (GI) abnormalities
10. Patients with non-healing wounds on any part of the body

Patients to be Excluded (patients must not meet any of the following criteria Phase 2a only)

1. Women who are pregnant or lactating. Women of child-bearing potential (WOCBP) and fertile men with WOCBP partner(s), not using and not willing to use a medically effective method of contraception.
2. Patients with known central nervous system (CNS) or leptomeningeal metastases, or spinal cord compression not controlled by prior surgery or radiotherapy, or patients with symptoms suggesting CNS involvement for which treatment is required
3. Patients with a malignancy other than EGFR-overexpressing triple negative breast cancer, squamous histology non-small cell lung cancer, or squamous cell carcinoma of the head and neck.
4. Patients with hematologic abnormalities at baseline
5. Patients with a significant cardiovascular disease or condition
6. Patients with a significant ocular disease or condition
7. Patients with a significant pulmonary disease or condition
8. History of pneumonia within 6 months prior to the first study drug administration
9. Patients with significant gastrointestinal (GI) abnormalities
10. Patients with non-healing wounds on any part of the body
11. Patients without measurable disease according to RECIST v1.1
12. Patients with an active second malignancy within the last 2 years prior to entry

Drugs and Other Treatments to be Excluded

1. Any antineoplastic agent for the primary malignancy (standard or investigational), without delayed toxicity, within 4 weeks, 5 plasma half-lives, or twice the duration of the biological effect, whichever is shortest, prior to first study drug administration and during study with the exception of: Nitrosoureas and nitrogen mustard within 6 weeks prior to first study drug administration and during study
2. Any other investigational treatments during study. This includes participation in any medical device or other therapeutic intervention clinical trials.
3. Radiotherapy for target lesions within 4 weeks prior to first study drug administration and during study
4. Herbal preparations or related over-the-counter (OTC) preparations/supplements containing herbal ingredients aimed at treating the underlying malignancy within 2 weeks prior to first study drug administration and during study
5. Strong inhibitors and/or inducers of cytochrome P450 (CYP) isoenzyme 3A4 within 2 weeks prior to first study drug administration and during study
6. Immunosuppressive or systemic hormonal therapy within 2 weeks prior to first study drug administration and during study.
7. Prophylactic use of hematopoietic growth factors within 1 week prior to first study drug administration and during Cycle 1 of study; thereafter prophylactic use of growth factors is allowed as clinically indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Lakhani, MD, Principal Investigator — START Midwest
Locations (10):
- United States (10):
  - Yale, New Haven, Connecticut
  - START Midwest, Grand Rapids, Michigan
  - The Tisch Cancer Institute-Mt. Sinai, New York, New York
  - Fox Chase, Philadelphia, Pennsylvania
  - Texas Oncology Midtown, Austin, Texas
  - Texas Oncology-Baylor -Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology McAllen, McAllen, Texas
  - Texas Oncology NE San Antonio, San Antonio, Texas
  - Texas Oncology Tyler, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AVID100 20 mg/m^2: Phase 1 Cohort 1: Participants were administered 20 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- AVID100 40 mg/m^2: Phase 1 Cohort 2: Participants were administered 40 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- AVID100 80 mg/m^2: Phase 1 Cohort 3: Participants were administered 80 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- AVID100 120 mg/m^2: Phase 1 Cohort 4: Participants were administered 120 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- AVID100 180 mg/m^2: Phase 1 Cohort 5: Participants were administered 180 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- AVID100 220 mg/m^2: Phase 1 Cohort 6: Participants were administered 220 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- AVID100 270 mg/m^2: Phase 1 Cohort 7: Participants were administered 270 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- Phase 2a Expansion: AVID100 220 mg/m^2: Participants from expanded populations of mTNBC, SCCHN, and Sq-NSCLC with documented EGFR expression received the maximum tolerated dose (MTD) determined in Phase 1, comprising AVID100 220 mg/m^2 administered every 3 weeks IV, for at least 1 cycle. Extended treatment was permitted for participants tolerating and benefiting from treatment.
Period: Overall Study
Arm/Group | AVID100 20 mg/m^2 | AVID100 40 mg/m^2 | AVID100 80 mg/m^2 | AVID100 120 mg/m^2 | AVID100 180 mg/m^2 | AVID100 220 mg/m^2 | AVID100 270 mg/m^2 | Phase 2a Expansion: AVID100 220 mg/m^2
Started | 1 | 1 | 3 | 3 | 3 | 6 | 7 | 25
Completed | 1 | 1 | 3 | 3 | 3 | 6 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 25
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Trial Termination | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants treated with at least 1 dose
Groups:
- AVID100 80 mg/m^2 Cohort 3: Phase 1 Cohort 3: Participants were administered 80 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- Total: Total of all reporting groups
Arm/Group | AVID100 20 mg/m^2 | AVID100 40 mg/m^2 | AVID100 80 mg/m^2 Cohort 3 | AVID100 120 mg/m^2 | AVID100 180 mg/m^2 | AVID100 220 mg/m^2 | AVID100 270 mg/m^2 | Phase 2a Expansion: AVID100 220 mg/m^2 | Total
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 6 | 7 | 25 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 2 | 3 | 3 | 4 | 3 | 16 | 32
  >=65 years | 0 | 1 | 1 | 0 | 0 | 2 | 4 | 9 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 2 | 2 | 4 | 5 | 10 | 24
  Male | 1 | 1 | 2 | 1 | 1 | 2 | 2 | 15 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 1 | 3 | 3 | 2 | 6 | 5 | 22 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 7
  White | 1 | 1 | 3 | 2 | 2 | 6 | 7 | 16 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Region of Enrollment [Number; unit: Participants]
  United States | 1 | 1 | 3 | 3 | 3 | 6 | 7 | 23 | 47
  Canada | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Dose Escalation: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs) in Cycle 1
Description: Any of the following toxicities, if judged to be associated with study, were considered a DLT:
  1. Evidence of pulmonary fibrosis
  2. G3 non-hematologic toxicity regardless of duration with the exceptions of:
     * G3 nausea, vomiting, diarrhea, or fatigue lasting < 2 days
     * G3 asymptomatic electrolyte abnormalities lasting < 3 days not considered clinically relevant
  3. AST and/or ALT elevation > 3 x ULN with total bilirubin > 2 x ULN without initial findings of cholestasis, that cannot be explained by other factors
  4. Any G4 non-hematologic toxicity with the exception of:
     • G4 asymptomatic electrolyte abnormalities lasting < 7 days not considered clinically significant
  5. Neutropenia that is:
     * > G3 and associated with fever
     * G4 and sustained (ANC < 500 per mm3, duration > 5 days)
  6. Thrombocytopenia that is:
     * G3 with clinically significant hemorrhage or requirement for transfusion
     * G4 (platelets < 25,000 per mm3)
  7. Inability to complete Cycle 1 at the assigned dose
Time Frame: Cycle 1 during Dose Escalation (ie the first 3 weeks of dosing)
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation Phase 1-Cohort 1: 1 Patient treated at 20mg/m2, AVID100 IV is administered once every 3 weeks
- Dose Escalation Phase 1-Cohort 2: 1 Patient treated at 40mg/m2, AVID100 IV is administered IV once every 3 weeks
- Dose Escalation Phase 1-Cohort 3: 3 Patients treated at 80mg/m2, AVID100 IV administered once every 3 weeks
- Dose Escalation Phase 1-Cohort 4: 3 Patients treated at 120mg/m2, AVID100 IV is administered once every 3 weeks
- Dose Escalation Phase 1-Cohort 5: 3 Patients treated at 180mg/m2, AVID100 IV is administered once every 3 weeks
- Dose Escalation Phase 1-Cohort 6: 6 Patients treated at 220 mg/m2, AVID100 IV is administered once every 3 weeks
- Dose Escalation Phase 1-Cohort 7: 7 Patients treated at 270mg/m2, AVID100 IV is administered once every 3 weeks
Arm/Group | Dose Escalation Phase 1-Cohort 1 | Dose Escalation Phase 1-Cohort 2 | Dose Escalation Phase 1-Cohort 3 | Dose Escalation Phase 1-Cohort 4 | Dose Escalation Phase 1-Cohort 5 | Dose Escalation Phase 1-Cohort 6 | Dose Escalation Phase 1-Cohort 7
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Phase 2a: Number of Participants With Best Overall Response by RECIST 1.1
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST 1.1 at Screening and every 2 cycles during study treatment.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non- target) must have reduction in short axis to < 10 mm.
Time Frame: Imaging for Disease status (tumour measurements) occurred after every even cycle for the full duration of treatment and at EOT visit up to approximately 24 weeks total
Population: Patients who completed Cycle 2 (6 weeks) of treatment, received at least 2 planned doses during that period, and had a follow-up assessment of disease status were considered evaluable for assessment of antineoplastic activity. Patients who were withdrawn from the study before completion of Cycle 2 because of progressive disease also were included in assessments of antineoplastic activity.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a Expansion: AVID100 220 mg/m^2
Number analyzed (Participants) | 24
Participants
  Progressive Disease | 23
  Stable Disease | 0
  Complete Response | 1

3. Secondary Outcome: PK Profile of Total Antibody
Description: Characterization of the pharmacokinetic profile of total antibody
Time Frame: Cycle 1 Profile (ie the first 3 weeks of dosing)
Population: Patients who have completed Cycle 1 for which PK analysis was performed
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- AVID100 40 mg/m^2: Phase 1 Cohort 1: Participants were administered 40 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- AVID100 80 mg/m^2: Phase 1 Cohort 1: Participants were administered 80 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- AVID100 120 mg/m^2: Phase 1 Cohort 1: Participants were administered 120 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- AVID100 180 mg/m^2: Phase 1 Cohort 1: Participants were administered 180 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- AVID100 220 mg/m^2: Phase 1 Cohort 1: Participants were administered 220 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
- AVID100 270 mg/m^2: Phase 1 Cohort 1: Participants were administered 270 mg/m^2 of AVID100 every 3 weeks, via intravenous catheter (IV), for a minimum of 1 cycle, with 1 month of follow-up after the last dose was administered.
Arm/Group | AVID100 20 mg/m^2 | AVID100 40 mg/m^2 | AVID100 80 mg/m^2 | AVID100 120 mg/m^2 | AVID100 180 mg/m^2 | AVID100 220 mg/m^2 | AVID100 270 mg/m^2 | Phase 2a Expansion: AVID100 220 mg/m^2
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 6 | 7 | 9
ng/mL
  Cycle 1 D1 prior SOI | NA — BLQ (below detection limit) | NA — BLQ (below detection limit) | NA (NA) — BLQ (below detection limit) | NA (NA) — BLQ (below detection limit) | NA (NA) — BLQ (below detection limit) | NA (NA) — BLQ (below detection limit) | NA (NA) — BLQ (below detection limit) | NA (NA) — BLQ (below detection limit)
  Cycle D1 EOI | 9213.3 | 13686.7 | 41140.7 (7472.0) | 71440.9 (9107.3) | 85982.9 (8517.2) | 113401.6 (18740.3) | 136306.3 (16938.5) | 122464.3 (20790.1)
  Cycle 1 D1 2h post SOI | 8066.3 | 14003.5 | 36935.8 (7089.3) | 66587.4 (6199.4) | 89676.6 (6216.5) | 112663.3 (21616.7) | 131267.2 (10585.7) | NA (NA) — Timepoint not assessed in Phase 2a expansion
  Cycle 1 D1 4h post SOI | 8351.9 | 14555.1 | 34399.7 (5940.6) | 61468.6 (4879.1) | 79581.1 (9542.3) | 101809.1 (17330.1) | 132671.4 (13243.3) | NA (NA) — Timepoint not assessed in Phase 2a expansion
  Cycle 1 D2 | 3217.6 | 9390.7 | 25236.4 (2159.3) | 43504.6 (5940.3) | 63001.5 (5837.3) | 68284.5 (6605.4) | 99382.8 (13832.9) | NA (NA) — Timepoint not assessed in Phase 2a expansion
  Cycle 1 D4 | 876.3 | 4578.3 | 14638.5 (1776.9) | 24985.3 (6859.7) | 35500.0 (5004.5) | 38068.0 (7890.3) | 69578.4 (10616.0) | NA (NA) — Timepoint not assessed in Phase 2a expansion
  Cycle 1 D8 | NA — BLQ (below detection limit) | NA — BLQ (below detection limit) | 2450.7 (1422.7) | 8768.0 (5393.1) | 12590.0 (1531.9) | 18581.5 (3128.7) | 27982.5 (13531.7) | NA (NA) — Timepoint not assessed in Phase 2a expansion
  Cycle 2 D1 prior to SOI | NA — BLQ (below detection limit) | NA — BLQ (below detection limit) | NA (NA) — BLQ (below detection limit) | NA (NA) — BLQ (below detection limit) | NA (NA) — BLQ (below detection limit) | NA (NA) — BLQ (below detection limit) | 866.5 (855.8) | 131.1 (40.6)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected after informed consent was signed for treatment and up to 30days following their last treatment or until an adverse event was as resolved up to approximately 28 weeks total.
Arm/Group | AVID100 20 mg/m^2 | AVID100 40 mg/m^2 | AVID100 80 mg/m^2 | AVID100 120 mg/m^2 | AVID100 180 mg/m^2 | AVID100 220 mg/m^2 | AVID100 270 mg/m^2 | Phase 2a Expansion: AVID100 220 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/3 | 0/3 | 0/3 | 0/6 | 1/7 | 3/25
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/3 | 2/3 | 1/3 | 3/6 | 2/7 | 13/25
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 3/3 | 3/3 | 6/6 | 7/7 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVID100 20 mg/m^2 (N=1) | AVID100 40 mg/m^2 (N=1) | AVID100 80 mg/m^2 (N=3) | AVID100 120 mg/m^2 (N=3) | AVID100 180 mg/m^2 (N=3) | AVID100 220 mg/m^2 (N=6) | AVID100 270 mg/m^2 (N=7) | Phase 2a Expansion: AVID100 220 mg/m^2 (N=25)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Progression of Disease (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Influenza A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension Crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper GI Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphasia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract Obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Super Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural hemorrhages (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AST increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
ALT increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uncontrolled pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet decrease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shortness of breath with hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatine Kinase increase (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multifocal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated AST (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVID100 20 mg/m^2 (N=1) | AVID100 40 mg/m^2 (N=1) | AVID100 80 mg/m^2 (N=3) | AVID100 120 mg/m^2 (N=3) | AVID100 180 mg/m^2 (N=3) | AVID100 220 mg/m^2 (N=6) | AVID100 270 mg/m^2 (N=7) | Phase 2a Expansion: AVID100 220 mg/m^2 (N=25)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 2 (2) | 4 (4) | 8 (8)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Conjunctivitis Allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Blood Alkaline Phosphate Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 1 (1) | 5 (12) — MedDRA 23.0 used for Phase 2
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (4) | 2 (3) | 6 (13) — MedDRA 23.0 for Phase 2
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 6 (7) — MedDRA 23.0 used for Phase 2
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 12 (16) — MedDRA 23.0 for Phase 2
Dermatitis Acneform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 5 (7)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperuricaemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — MedDRA 23.0 for Phase 2
Dysphagia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) — MedDRA 23.0 for Phase 2 event
Face Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 23.0 for Phase 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — MedDRA 23.0 for Phase 2
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) — MedDRA 23.0 for Phase 2
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — MedDRA 23.0 for Phase 2
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — MedDRA 23.0 for Phase 2
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — MedDRA 23.0 for Phase 2
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Alkaline Phosphatase Increase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Anorexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT03094169/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT03094169/ICF_001.pdf